CLINICAL TRIAL: NCT05912946
Title: Assessing the Effectiveness and Safety of Interferon Bladder Infusion for the Treatment of Interstitial Cystitis: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Assessing the Effectiveness and Safety of Interferon Bladder Infusion for the Treatment of Interstitial Cystitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, De-yi Luo, Prof, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022370
Record Dates: First submitted 2023-05-30; First posted 2023-06-22 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Interstitial Cystitis
Keywords: Interstitial cystitis; Interferon; Bladder infusion
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Interferons; Hyaluronic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group drug (Experimental): Generic name: Human interferon a2b injection; Dosage form: solution; Dosage: 1ml: 3 million IU; Frequency and duration: The first 4 weeks were irrigated once a week, a total of 4 times, and the last 4 months were irrigated once a month, a total of 4 times. The total treatment cycle was 5 months, and a total of 8 bladder perfusion treatments were performed.
  Interventions: Drug: Interferon
- Sodium Hyaluronate (Active Comparator): Generic name: Sterile sodium hyaluronate solution; Dosage form: solution; Dosage: 40mg/50ml; Frequency and duration: The first 4 weeks were irrigated once a week, a total of 4 times, and the last 4 months were irrigated once a month, a total of 4 times. The total treatment cycle was 5 months, and a total of 8 bladder perfusion treatments were performed.
  Interventions: Drug: Sodium Hyaluronate
- Sodium chloride injection (Placebo Comparator): Generic name: Sodium chloride injection; Dosage form: solution; Dosage: 50ml: 0.45g; Frequency and duration: The first 4 weeks were irrigated once a week, a total of 4 times, and the last 4 months were irrigated once a month, a total of 4 times. The total treatment cycle was 5 months, and a total of 8 bladder perfusion treatments were performed.
  Interventions: Drug: Sodium Chloride Injection

INTERVENTIONS:
Drug: Interferon — The patient was seated in the seat and rested quietly. A three-way urinary tube was indwelled to drain urine. Interferon solution was configured according to the ratio of 3 million IU interferon +49ml normal saline. The urinary tube was clamped and the interferon solution was injected through the water inlet tube and retained for 30 minutes.
  Arms: Experimental group drug
Drug: Sodium Hyaluronate — The patient was seated in the seat and rested quietly. A three-way urinary tube was indwelled to drain urine. The urinary tube was clamped and the sterile sodium hyaluronate solution was injected through the water inlet tube and retained for 30 minutes.
  Arms: Sodium Hyaluronate
Drug: Sodium Chloride Injection — The patient was seated in the seat and rested quietly. A three-way urinary tube was indwelled to drain urine. The urinary tube was clamped and the sodium chloride injection was injected through the water inlet tube and retained for 30 minutes.
  Arms: Sodium chloride injection

SUMMARY:
Interstitial cystitis/bladder pain syndrome (IC/BPS) is one of the most intractable diseases of Urogynecology. The main clinical manifestations of interstitial cystitis/bladder pain are frequent urination and severe overflowing bladder pain. Due to the unclear pathological mechanism and the diversity of clinical manifestations and pathological features of the disease, the diagnosis is mainly to exclude suspicious diseases. At present, IC/BPS treatment mainly includes oral administration of mast cell stabilizing drugs such as sodium pentosan sulfate and anticholinergic drugs, or bladder instillation of dimethyl sulfone, hyaluronic acid and other drugs directly acting on the bladder mucosa, or surgical treatment such as sacrospinal radiculotomy and peripheral denervation of the bladder, but all can only relieve clinical symptoms and improve quality of life, and can not be targeted etiological treatment according to the pathological mechanism. Research showed JC polyomavirus (JCPyV) virus may be the original pathogen causing the development of IC/BPS. Interferon, as a broad-body antiviral agent, plays a critical role in triggering innate and adaptive immune responses against viral replication and infection. It can inhibit the replication and transcription of JCPyV through a variety of pathways. Interferon may be a potential specific drug for IC/BPS. Therefore, this study aims to evaluate the efficacy and safety of interferon bladder perfusion for IC/BPS.

DETAILED DESCRIPTION:
The main manifestations of IC/BPS patients are pain, pressure or discomfort related to the bladder. Due to the unclear pathogenesis and inconsistent diagnostic criteria, accurate and effective clinical diagnosis and treatment of IC/BPS become very difficult. The diagnosis of IC/BPS is often uncertain and delayed, with patients moving from one hospital to another, often taking 2-11 years to get a final diagnosis. At present, the treatment of IC/BPS is mostly aimed at relieving clinical symptoms (including drugs, bladder perfusion, sacral nerve regulation, etc.), instead of radical treatment based on pathological mechanism. However, the long-term follow-up effect of commonly used clinical treatment is not good, with a recurrence rate of 70%. And about 10% of patients will eventually choose bladder resection because of the physical torture and mental stress caused by the disease. Previous studies confirmed that the positive rate of JCPyV in the urine of IC/BPS patients was 95%, while no JCPYV was found in the control group, suggesting that JCPYV may play an important role in the pathological mechanism of IC/BPS. The literature review also confirmed the presence of BK polyomaviruses (BKPyV) and JCPyV in IC/BPS urine, and a case of bladder perfusion therapy with interferon was reported to alleviate the frequency of urination and pain symptoms in IC/BPS patients, suggesting that interferon may be a potential specific drug for IC/BPS treatment. However, there are basically no relevant clinical studies at present. Therefore, this study aims to explore the efficacy and safety of interferon intravesical infusion therapy for IC/BPS. The research results are expected to improve the existing therapeutic means and explore new therapeutic targets. It lays an important foundation for the accurate treatment of IC/BPS.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old, regardless of gender
* Combined with bladder pain/discomfort during urination, and at least one lower urinary tract symptom such as frequency and urgency, duration > 6 months
* The total score of O'Leary-Sant ICSI+ICPI is more than 18 points
* Agree to receive bladder perfusion therapy

Exclusion Criteria:

* Have a history of allergy to interferon drugs
* Patients with serious heart, lung, liver, kidney or blood diseases, abnormal liver function, renal insufficiency, etc.
* Pregnant or lactating women
* A history of urinary tract infection within 12 weeks
* IC/ BPS-like symptoms caused by urinary diseases, such as overactive bladder, neurogenic bladder, urinary calculi, radiation cystitis, and endometriosis
* Within 24 weeks, patients had the following treatment history: bladder hydrodilation, intravesical laser treatment, pelvic floor reconstruction surgery
* Patients who have taken related drugs or participated in other clinical studies and received study drugs or medical device interventions within 3 months

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
The score of global response assessment (GRA) pre- and post-treatment | The time frame was from the date of bladder infusion to the date of final follow-up, ranging from 1 to 12 months
  The primary treatment outcomes were assessed using the Global Response Assessment (GRA) score (categorized into - 3, - 2, - 1, 0, 1, 2, and 3, indicating markedly worse to markedly improved status)
The score of visual analogue scale (VAS) pre- and post-treatment | The time frame was from the date of bladder infusion to the date of final follow-up, ranging from 1 to 12 months
  The score of VAS ranging from 0 to 10. Higher scores indicate higher levels of pain.
Interstitial Cystitis Symptom Average Index (ICSI) questionnaires pre- and post-treatment | The time frame was from the date of bladder infusion to the date of final follow-up, ranging from 1 to 12 months
  The O'Leary-Sant instrument is comprised of Symptom Index (score range: 0-20 points), which contains four questions related to urinary and pain symptoms.
  The score is calculated by summing the points for each item, and a score ≥6 points indicates IC.
Interstitial Cystitis Problem Average Index (ICPI) questionnaires pre- and post-treatment | The time frame was from the date of bladder infusion to the date of final follow-up, ranging from 1 to 12 months
  The O'Leary-Sant instrument is comprised of Problem Index (score range: 0-16 points), which contains four questions related to urinary and pain symptoms.
  The score is calculated by summing the points for each item, and a score ≥6 points indicates IC.
The score of pelvic pain and urgency/frequency (PUF) pre- and post-treatment | The time frame was from the date of bladder infusion to the date of final follow-up, ranging from 1 to 12 months
  The score ranges from 0 to 35 points. A score ≥5 points is considered to indicate IC.

SECONDARY OUTCOMES:
Treatment-related complications | The time frame was from the date of bladder infusion to the date of final follow-up, ranging from 1 to 12 months
  Treatment-related complications, such as urinary tract infections, pain, psychiatric symptoms, changes in liver and kidney function, and gastrointestinal symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-min Li, Study Chair — West China Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shen SH, Peng L, Zeng X, Zhang J, Shen H, Luo DY. Intravesical Interferon Therapy vs Hyaluronic Acid for Pain Among Female Individuals With Interstitial Cystitis: A Randomized Clinical Trial. JAMA Netw Open. 2024 Apr 1;7(4):e244880. doi: 10.1001/jamanetworkopen.2024.4880. PMID 38587846